CLINICAL TRIAL: NCT05473416
Title: Comparing the Effects of Pilates (Pelvic Tilt) and McKenzie Back Extension Exercises in Power Loom Workers Having Non-specific Chronic Low Back Pain
Brief Title: Comparing the Effects of Pilates and McKenzie in Power Looms Workers Having Nonspecific Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, HAFIZ MUHAMMAD ALMAS SABIR, Principle Investigator, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAFIZ MUHAMMAD ALMAS SABIR
Record Dates: First submitted 2022-07-18; First posted 2022-07-25 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Nonspecific Chronic Low Back Pain; Pain; Disability Physical
Keywords: Pilates pelvic tilt exercise & McKenzie back exercise
MeSH Terms: conditions — Pain | interventions — RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: The study was based on the research design of a randomized clinical trial. The single-blind study, in which participants were blind. The sample size of this study was 46. Patient was divided into 2 groups, 23 in each group.
Who Masked: Participant
Masking Description: participants were blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1- McKenzie (Group A) (Experimental): Back extension exercise. Total 10 repetitions in 1 set. Total 3 sets in a session. Total 3 sessions in a week. Total 12 sessions in a month.
  Interventions: Other: McKenzie back extension exercise; Other: Baseline treatment
- 2- Pilates (Group B) (Experimental): Pelvic tilt exercise Total 10 repetitions in 1 set. Total 3 sets in a session. Total 3 sessions in a week. Total 12 sessions in a month.
  Interventions: Other: Pilates pelvic tilt exercise; Other: Baseline treatment

INTERVENTIONS:
Other: McKenzie back extension exercise — McKenzie's back extension exercise consists; start with your belly facing down on the mat. Angle your legs in line with your hips, point your toes, and breathe into the next movement. Gently bending your elbows, push yourself up off the floor, until you feel the extension in your back. Be mindful not to lock your elbows as you support your weight with your hands and wrists for 10 seconds. Take deep inhales and exhales as you move in and out of the pose. Patients will be performed these activities under the supervision of physiotherapist.
  Arms: 1- McKenzie (Group A)
Other: Pilates pelvic tilt exercise — Pilates pelvic tilt exercise consists; lie with your back on the floor in a neutral position with your legs bent and toes facing forward. Pull your belly button in toward your spine, pushing your pelvis up toward the ceiling. Tighten your gluteus and hip muscles as you tilt your pelvis forward. Hold for 10 seconds.
  Arms: 2- Pilates (Group B)
Other: Baseline treatment — Postural guidelines + proper lifting technique + stretch break Rest
  Other Names: Postural guidelines + stretch break + rest

SUMMARY:
to check the effects of Mckenzie intervention & Pilates intervention on power looms workers having nonspecific chronic low back pain

DETAILED DESCRIPTION:
The purpose of this study is to check and compare the effects of McKenzie back extension exercise and Pilates pelvic tilt exercise on power looms workers having nonspecific chronic low back pain. To check the effects of these interventions on pain, disability, and anterior pelvic tilt angle.

In this study pain intensity of the subjects will be noted via a numeric pain rating scale. Pain will be measured at baseline, after 2 weeks and 4 weeks of intervention.

In this study disability of the patients will be measured via Quebec back pain disability scale. Disability will be measured at baseline, after 2 weeks and 4 weeks of intervention.

In this study, a goniometer will be used to measure the anterior pelvic tilt angle. Anterior pelvic tilt angle will be measured at baseline, after 2 weeks and 4 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age of the participants between 35-45 years.
* Only male workers diagnosed with nonspecific chronic low back pain.
* Power looms workers; Operator of power looms, working 12 hours per day.
* Low back pain for more than three months.
* Power looms workers with pain intensity on NPRS ranges from mild to moderate.
* Anterior pelvic tilt angle more than normal 13º±4.9º, anteriorly tilt to 18º to 25º.

Exclusion Criteria:

* Serious spinal pathology like tumors.
* Any inflammatory diseases.
* History of spinal surgery.
* Neurological disorder.
* Pain due to any systemic diseases.

Ages: 35 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only Male
Enrollment: 46 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-11-13 (Actual); Study Completion 2022-12-24 (Actual)

PRIMARY OUTCOMES:
Pain intensity | one month
  In this study pain intensity of the subjects will be noted via numeric pain rating scale. The reading of NPRS is in number from 0 to 10 where 0 mean no pain, 10 means worst pain, 1-3 indicate mild pain, 4-6 present moderate pain, and 7-10 means severe pain. Patient tell us in numeric form how much he feels pain for example patient tell us he has 4 pain; its mean patient has moderate pain.
Disability index | one month
  In this study disability of the patients will be measured via Quebec back pain disability scale. The 20-item Quebec back pain Disability Scale for Back Pain was created to measure degree of functional disability in people who have low back pain. The scale is a dependable and valid measurement used to evaluate each patient's improvement during treatment or rehabilitation programmers.

SECONDARY OUTCOMES:
Anterior pelvic tilt angle abnormailty | one month
  In this study goniometer was used to measure the anterior pelvic tilt angle of the power loom workers. Goniometer has three parts the body, stationary arm, and the mobile arm. To check the anterior pelvic tilt angle in subjects the body of the goniometer was placed on the anterior superior iliac spine horizontally, mobile arm was moved to the posterior superior iliac spine and noted the reading displayed on the goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiz Muhammad Almas Sabir Muhammad Sabir Ali, MS OMPT, Principal Investigator — The University of Faisalabad
Locations (1):
- Dr Hafiz Almas PT, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No